CLINICAL TRIAL: NCT03294525
Title: Clinical Psychopharmacology Division
Brief Title: Towards Neurobiology-based Diagnosis and Treatment of Affective Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Clinical Psychopharmacology Division, Peking University
Other Study IDs: 001
Record Dates: First submitted 2016-05-24; First posted 2017-09-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Affective Disorder
MeSH Terms: conditions — Mood Disorders | interventions — Escitalopram; Duloxetine Hydrochloride; Mirtazapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected by venepuncture.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Escitalopram-for MDD: Eligible patients were assigned to escitalopram treatment based on investigators' clinical practice.
  Interventions: Drug: Escitalopram Pill
- Duloxetine-for MDD: Eligible patients were assigned to duloxetine treatment based on investigators' clinical practice.
  Interventions: Drug: Duloxetine
- Mirtazepine-for MDD: Eligible patients were assigned to mirtazepine treatment based on investigators' clinical practice.
  Interventions: Drug: Mirtazapine Pill
- other antidepressant-for MDD: Eligible patients were assigned to other antidepressant treatment (including sertraline, paroxetine, fluoxetine, venlafaxine, etc) based on investigators' clinical practice.
  Interventions: Drug: Other Antidepressants

INTERVENTIONS:
Drug: Escitalopram Pill — escitalopram 10~20mg/day
  Other Names: Lexapro
  Groups: Escitalopram-for MDD
Drug: Duloxetine — duloxetine 30~120mg/day
  Other Names: Cymbalta
  Groups: Duloxetine-for MDD
Drug: Mirtazapine Pill — Mirtazapine 15~45mg/day
  Other Names: Remeron
  Groups: Mirtazepine-for MDD
Drug: Other Antidepressants
  Groups: other antidepressant-for MDD

SUMMARY:
The project is a multi-center, prospective cohort study. The study's total targeted enrollment is 400 first-episode patients with major depressive disorder (MDD) and 400 healthy controls.

DETAILED DESCRIPTION:
Four hundred patients with a primary diagnosis of depression and HAMD-17 scores ≥14 at baseline visit are to be assigned to one of the second-generation antidepressant drugs, including escitalopram, duloxetine, mirtazapine, paroxetine, sertraline, etc based on investigators' clinical practice. Initial treatment consists of a 8-week course with one of these monotherapies. Patients who meet criteria for full remission are followed for a 22-month follow-up phase to monitor for depression recurrence. Patients who do not remit are offered another 8 weeks of acute treatment, including combination therapy or switching to other antidepressant based on investigators' clinical practice. The clinical assessment (Hamilton Depression Rating Scale(HAMD)/ Clinical general impression (CGI) /the Positive and Negative Affect Schedule (PANAS) /subtypes of depression, Dimensional Anhedonia Rating Scale (DARS) , etc), early life stress, neuropsychological test, and biological examination (MRI, genetics, neurochemistry, and immunology) were conducted to identify the biomarkers associated with diagnosis, treatment efficacy prediction of depression. Among the 400 patients, about 100 patients receive MRI scans at baseline and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with depression

* The inclusion criteria for depressed patients were: male or female outpatients aged between 18 and 55 years old
* Currently in acute depressive episode
* Total HAMD-17 score≥14 at baseline visit.
* The diagnosis of depression was confirmed by a trained psychiatrists using the Mini-International Neuropsychiatric Interview (MINI).
* The patients participating in imaging scans should additionally satisfy: not taking psychiatric drugs within last two weeks (except for benzodiazepine) or fluoxetine last one month
* Not receiving ECT within last 6 months.

Exclusion Criteria:

* Unable to complete the questionnaire and psychological assessment independently
* Significant cognitive impairments determined by system mental examination and inability to sign an informed consent form
* Past or presently suffering from other psychiatric disorders, alcohol and drug dependence
* Suffering from major physical diseases, such as cardiovascular and cerebrovascular diseases, respiratory diseases, kidney disease, cancer and so on; personality disorder
* Intellectual disabilities
* Suicidal behavior
* Being participating in other studies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with major depressive disorder
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
reduction in HAMD total scores | 8 weeks
  reduction more than 50% was regarded as response
remision | 8 weeks
  HAMD total score less than 7

CONTACTS AND LOCATIONS:
Overall Officials: Tianmei Si, PhD, Principal Investigator — Sixth hospital of beijing university
Locations (1):
- Institute of mental health, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai YR, Wu YK, Chen X, Zeng YW, Li K, Li JT, Su YA, Zhu LL, Yan CG, Si TM. Eight-week antidepressant treatment changes intrinsic functional brain topology in first-episode drug-naive patients with major depressive disorder. J Affect Disord. 2023 May 15;329:225-234. doi: 10.1016/j.jad.2023.02.126. Epub 2023 Feb 28. PMID 36858265
- [Derived] Lin J, Su Y, Rizvi SJ, Jagoda J, Li J, Wu Y, Dai Y, Zhang Y, Kennedy SH, Si T. Define and characterize the anhedonia in major depressive disorder: An explorative study. J Affect Disord. 2022 Sep 15;313:235-242. doi: 10.1016/j.jad.2022.06.082. Epub 2022 Jul 3. PMID 35788366
- [Derived] Li L, Su YA, Wu YK, Castellanos FX, Li K, Li JT, Si TM, Yan CG. Eight-week antidepressant treatment reduces functional connectivity in first-episode drug-naive patients with major depressive disorder. Hum Brain Mapp. 2021 Jun 1;42(8):2593-2605. doi: 10.1002/hbm.25391. Epub 2021 Feb 27. PMID 33638263